CLINICAL TRIAL: NCT01915654
Title: Impact de la Transfusion de Culots Globulaires de Moins de 14 Jours Sur la Morbi-mortalité Chez Des Patients en Chirurgie Cardiaque
Brief Title: Impact of RBC Transfusion Less Than 14 Days on Morbidity and Mortality in Cardiac Surgical Patients
Acronym: CGRCard
Status: Terminated | Type: Observational
Why Stopped: Retrospective study from December 2007 to May 2010
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/194
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery; Transfusion Related Complication
Keywords: Cardiac surgery; Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study population: The study involves patients operated in the cardiothoracic and cardio-vascular surgery department of Besançon University Hospital between December 2008 and May 2009 (study population) or between December 2007 and May 2008 and between December 2009 and May 2010 (reference population).
  Interventions: Procedure: study population
- Reference population: The study involves patients operated in the cardiothoracic and cardio-vascular surgery department of Besançon University Hospital between December 2008 and May 2009 (study population) or between December 2007 and May 2008 and between December 2009 and May 2010 (reference population).

INTERVENTIONS:
Procedure: study population — Population of patients undergoing cardiac surgery between December 2008 and May 2009, with pellets transfused RBCs stored for less than 14 days
  Groups: Study population

SUMMARY:
The purpose of the transfusion of packed red blood cell is to overcome acute or chronic anemia cause tissue hypoxia. It increases hemoglobin concentration and consequently increase oxygen delivery to peripheral tissues. The perioperative period of major surgery is a field particularly favorable to the development of tissue hypoxia, which is associated with increased mortality and postoperative morbidity. Optimization of oxygen transport to tissues at the preoperative period is accompanied by a significant reduction of these major complications.

Clinical complications (infectious or otherwise) related to transfusion of caps Red Blood cells Caps (RBC)are well known. Many studies seem to evidence the potentially deleterious effect of transfusion, especially in patients with poor condition, related to storage time. Indeed, during storage, impaired blood-related storage is created. It is metabolic, biochemical and molecular levels. Many studies, carried out in particular in cardiac surgery where patients are suitable for transfusion RBC, have focused on the effect of transfusions on consumption and the transport of oxygen to demonstrate the impact of conservation lesions on their role in vivo. In particular, a single-center retrospective American study showed reduction of postoperative complications in patients who received RBC under 14 days.

However one of the confounding factors present is that all transfused RBCs are not leukoreduced (unlike the French transfusion policy). In addition, the greater part of the clinical studies are controversial. That is why we aim to assess, through a retrospective study of data, the impact of transfusion of red red blood cells within 14 days of post-operative morbidity and mortality, compared to the usual transfusion practice in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients male or female over the age of 18 years
* Patients able to understand the benefits and risks of testing
* For the study population: patients who underwent cardiac surgery (all surgery combined) scheduled or emergency December 2008 to May 2009, having been transfused intraoperatively and until the seventh postoperative day .
* For the reference population: patients who have undergone elective or emergency cardiac surgery from December 2007 to May 2008 and from December 2009 to May 2010, having been transfused intraoperatively and until the seventh postoperative day.

Exclusion Criteria:

* Inability to understand the advantages and disadvantages of the study, psychiatric disorders judged by the investigator to be incompatible with the inclusion in the study.
* Patients who have expressed opposition to his participation in the study.
* For the study population: patients were transfused within seven days before the start of the observation period.
* For the study population: patients with transfusion of red blood cell more than 14 days
* For the reference population: patients were transfused within seven days before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves patients operated in the cardiothoracic and ardio-vascular surgery department of Besançon University Hospital between December 2008 and May 2009 (study population) or from December 2007 to May 2008 and from December 2009 to May 2010 (reference population).
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
death / acute renal failure / operating / stroke / postoperative ischemia post infection | in-beyond the 48th hour of the transfusion
  The primary endpoint was the occurrence of death and / or acute renal failure and / or operating and / or stroke and / or postoperative ischemia post infection, in-beyond the 48th hour of the transfusion.

SECONDARY OUTCOMES:
Mortality / average length of stay in intensive care / resuscitation (> 48 hours) / the average length of stay in cardiac surgery | 30 days
  The secondary endpoints were mortality at 30 days, the average length of stay in intensive care / resuscitation (> 48 hours) and (> 15 days).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Flicoteaux, Principal Investigator — CHRU de Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France, France